CLINICAL TRIAL: NCT05345652
Title: Evaluation Of Deep Anterior Lamellar Keratoplasty By Anterior Segment Ocular Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Omar Mohamed Ali, Principal Investigator, Assiut University
Other Study IDs: Ant. segment OCT in DALK
Record Dates: First submitted 2022-03-29; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Keratoconus; Cornea; Corneal Opacity
MeSH Terms: conditions — Keratoconus; Corneal Diseases; Corneal Opacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: deep anterior lamellar keratoplasty — DALK is a partial-thickness corneal transplant which involves only the donor stroma, leaving the recipient's own Descemet's membrane and endothelium
  Other Names: DALK

SUMMARY:
Investigators' research is concerned observing the post-operative anterior segment OCT changes throughout the post- operative follow up of the patient and relating to improve the visual outcome of the surgery which is the goal of surgery

DETAILED DESCRIPTION:
Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):

* Complete medical and ocular history, including patients' age, sex, type of pathology of the cornea such as keratoconus, opacity , history of previous corneal intervention , and other ocular surgeries.
* Thorough ophthalmological examination, including visual acuity, intraocular pressure (IOP) measuring by Goldman applanation tonometer (Haag Streit, Koeniz, Switzerland), slit lamp biomicroscopic examination of anterior segment, investigations for keratoconus as pentacam , preoperative anterior segment OCT if needed , slit lamp photography for the cornea .

Candidate patients will be operated through DALK , then will be examined post operative clinically and be followed up at 3 months , 6 months for best corrected visual acuity, Intraocular pressure , refraction , graft healing , and anterior segment OCT for the anterior chamber angel , graft healing , descemet's membrane state , tear film . The interpretation of the clinical data with the changes in the ant. Segment OCT will give us the clue to get the best visual outcome of surgery .

2.4.5 -Research outcome measures:

1. Primary (main):

   To evaluate the post-operative changes after DALK surgery through ant segment OCT and its relation to clinical findings.
2. Secondary (subsidiary): To improve the outcome of the surgery through the graft creation , stitching of the graft , following up the IOP clinically and state of AC angel through OCT , the tear film and changes after surgery , all these factors to improve the target of the surgery which is the post operative best corrected visual acuity .

Data collection Data to be collected include patients' age, sex, cause of corneal surgery ,BCVA, IOP levels, clinical examination of the eye and if there are findings , and ant. Segment OCT of the eye Computer software Data analysis will be done via SPSS version 26 windows 10 Statistical tests Data will be statistically described in terms of mean, SD, and range when appropriate. Comparisons between the preoperative and postoperative data will be done using Student's t-test. Study groups' comparisons will be done using Student's t-test for independent normally distributed samples data.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing DALK surgery older than 18 years old ( keratoconus and corneal opacity ).

Exclusion Criteria:

* Patients suffering from active corneal ulcer
* Active infection.
* Posterior segment diseases.
* Recent ocular surgery in the study eye in the 2 months prior to enrolment,
* Media opacities as vitreous haemorrhage,
* Vasculitis , patients with macular edema related to, glaucoma, chronic uveitis, or pre-existing ocular pathologic features or abnormalities.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Older than 18 years old and younger than 60 in need for dalk
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-09-29 (Estimated)

PRIMARY OUTCOMES:
To evaluate the post-operative changes after DALK surgery through ant segment OCT and its relation to clinical findings. | 6 months after the surgery
  To evaluate the post-operative changes after DALK surgery through ant segment OCT and its relation to clinical findings.

SECONDARY OUTCOMES:
To Improve sugery | 6 months after the surgery
  To improve the post operative best corrected visual acuity .

CONTACTS AND LOCATIONS:
Overall Officials: momen A Mohammad, Lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hos D, Matthaei M, Bock F, Maruyama K, Notara M, Clahsen T, Hou Y, Le VNH, Salabarria AC, Horstmann J, Bachmann BO, Cursiefen C. Immune reactions after modern lamellar (DALK, DSAEK, DMEK) versus conventional penetrating corneal transplantation. Prog Retin Eye Res. 2019 Nov;73:100768. doi: 10.1016/j.preteyeres.2019.07.001. Epub 2019 Jul 3. PMID 31279005
- [Background] Singh R, Gupta N, Vanathi M, Tandon R. Corneal transplantation in the modern era. Indian J Med Res. 2019 Jul;150(1):7-22. doi: 10.4103/ijmr.IJMR_141_19. PMID 31571625
- [Result] Krumeich JH, Knulle A, Krumeich BM. [Deep anterior lamellar (DALK) vs. penetrating keratoplasty (PKP): a clinical and statistical analysis]. Klin Monbl Augenheilkd. 2008 Jul;225(7):637-48. doi: 10.1055/s-2008-1027485. German. PMID 18642207
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/31571625/